CLINICAL TRIAL: NCT02852278
Title: A Patient Centric Motor Neuron Disease Activities of Daily Living Scale
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Kansas (Other); University of Miami (Other)
Responsible Party: Sponsor
Other Study IDs: CReATe 8003; U01TR001263 (NIH)
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Amyotrophic Lateral Sclerosis; Progressive Muscular Atrophy; Primary Lateral Sclerosis; Hereditary Spastic Paraplegia
Keywords: Amyotrophic Lateral Sclerosis; ALS; motor neuron diseases; Progressive Muscular Atrophy; Primary Lateral Sclerosis; Hereditary Spastic Paraplegia
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Muscular Atrophy, Spinal; Motor Neuron Disease; Spastic Paraplegia, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Web-based Survey — This is a prospective 12-month study of patients with motor neuron disease enrolled in CReATe Connect, an RDCRN Contact Registry.

SUMMARY:
The purpose of this study is to learn about rates of patient-reported disease progression in patients with motor neuron diseases (amyotrophic lateral sclerosis, progressive muscular atrophy, primary lateral sclerosis, hereditary spastic paraplegia) outside the clinical setting, and the patient-reported clinical characteristics that influence this rate of progression. All patients enrolled in CReATe Connect, a Rare Diseases Clinical Research Network (RDCRN) Contact Registry, will be invited via email to participate in this study.

DETAILED DESCRIPTION:
The patient activities of daily living for amyotrophic lateral sclerosis survey (PADL-ALS, Appendix B) is a patient-centric revision of the standard revised ALS functional rating scale used in clinical trials, the ALSFRS-R. The PADL-ALS was developed based on patient interviews, and patient focus groups. The ALSFRS-R is made up of 12 categories detailing various activities of daily living and includes six bulbar-respiratory functions, three upper extremity functions (writing, cutting food, and dressing), and three gross motor functions (walking, climbing, and turning in bed). Each activity is recorded to the closest approximation from a list of five choices, scored 0-4, with the total score ranging from 48 (normal function) to 0 (no function). The PADL-ALS includes questions from the ALSFRS-R, with revisions to make the questions easier to understand. In addition the PADL-ALS contains a question about pain; a question about emotional lability; and a general non-denominational question about faith. The survey will be composed of two parts, the initial survey, and then monthly follow up surveys. The initial survey will include the PADL-ALS with additional questions about symptom onset, date of diagnosis, initial region involved, patient impression of diagnosis, general demographic questions (age, gender, race, ethnicity, education), and medications related to their diagnosis of motor neuron disease.

The survey data will be stored by the Rare Diseases Clinical Research Network's Data Management and Coordinating Center (DMCC) at the University of South Florida. Upon conclusion of the study period, the data will be sent to Jeffrey Statland, MD, University of Kansas Medical Center (Study Chair) and Michael Benatar, MD, PhD, University of Miami (CReATe Consortium PI). All data collected will be sent to the database of Genotypes and Phenotypes (dbGaP) to be stored indefinitely.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported diagnosis of motor neuron disease (amyotrophic lateral sclerosis, amyotrophic lateral sclerosis - frontotemporal dementia, primary lateral sclerosis, progressive muscular atrophy, or hereditary spastic paraplegia)
* Enrolled in CReATe Connect, an RDCRN Contact Registry

  o Individuals of any age, race, ethnicity, and from any location will be able to participate
* Participants will need to be able to fill out the survey in English

Exclusion Criteria:

• Inability to provide informed consent and complete survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with motor neuron disease enrolled in CReATe Connect, an RDCRN Contact Registry
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
PADL-ALS Survey | 12 months
  The PADL-ALS survey is a revision of the ALSFR-R, which consists of 12 categories detailing various activities of daily living and includes six bulbar-respiratory functions, three upper extremity functions (writing, cutting food, and dressing) and three gross motor functions (walking, climbing, and turning in bed). Each activity is recorded from a list of five choices, scored 0-4, with the total score ranging from 48 (normal function) to 0 (no function). The PADL-ALS includes questions from the ALSFRS-R, with revisions for easier understanding. The PADL-ALS also includes questions about pain, emotional lability and a general non-denominational question about faith. The survey is composed of an initial survey and monthly follow up surveys. The initial survey will include additional questions about symptom onset, date of diagnosis, initial region involved, patient impression of diagnosis, general demographic questions, and medications related to their diagnosis of motor neuron disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Statland, MD, Principal Investigator — University of Kansas Medical Center; Michael Benatar, MD, PhD, Principal Investigator — University of Miami; Jeffery Krischer, PhD, Principal Investigator — University of South Florida, Data Management Coordinating Center; Callyn Kirk, MSPH, Principal Investigator — University of South Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847
- [Background] Brooks BR. El Escorial World Federation of Neurology criteria for the diagnosis of amyotrophic lateral sclerosis. Subcommittee on Motor Neuron Diseases/Amyotrophic Lateral Sclerosis of the World Federation of Neurology Research Group on Neuromuscular Diseases and the El Escorial "Clinical limits of amyotrophic lateral sclerosis" workshop contributors. J Neurol Sci. 1994 Jul;124 Suppl:96-107. doi: 10.1016/0022-510x(94)90191-0. No abstract available. PMID 7807156
- [Result] Norris F, Shepherd R, Denys E, U K, Mukai E, Elias L, Holden D, Norris H. Onset, natural history and outcome in idiopathic adult motor neuron disease. J Neurol Sci. 1993 Aug;118(1):48-55. doi: 10.1016/0022-510x(93)90245-t. PMID 8229050
- [Result] Eisen A, Schulzer M, MacNeil M, Pant B, Mak E. Duration of amyotrophic lateral sclerosis is age dependent. Muscle Nerve. 1993 Jan;16(1):27-32. doi: 10.1002/mus.880160107. PMID 8423829
- [Result] Gubbay SS, Kahana E, Zilber N, Cooper G, Pintov S, Leibowitz Y. Amyotrophic lateral sclerosis. A study of its presentation and prognosis. J Neurol. 1985;232(5):295-300. doi: 10.1007/BF00313868. PMID 4056836
- [Result] The Amyotrophic Lateral Sclerosis Functional Rating Scale. Assessment of activities of daily living in patients with amyotrophic lateral sclerosis. The ALS CNTF treatment study (ACTS) phase I-II Study Group. Arch Neurol. 1996 Feb;53(2):141-7. PMID 8639063
- [Result] Bensimon G, Lacomblez L, Meininger V. A controlled trial of riluzole in amyotrophic lateral sclerosis. ALS/Riluzole Study Group. N Engl J Med. 1994 Mar 3;330(9):585-91. doi: 10.1056/NEJM199403033300901. PMID 8302340
- [Result] Miller RG, Bouchard JP, Duquette P, Eisen A, Gelinas D, Harati Y, Munsat TL, Powe L, Rothstein J, Salzman P, Sufit RL. Clinical trials of riluzole in patients with ALS. ALS/Riluzole Study Group-II. Neurology. 1996 Oct;47(4 Suppl 2):S86-90; discussion S90-2. doi: 10.1212/wnl.47.4_suppl_2.86s. PMID 8858057
- [Result] Cedarbaum JM, Stambler N, Malta E, Fuller C, Hilt D, Thurmond B, Nakanishi A. The ALSFRS-R: a revised ALS functional rating scale that incorporates assessments of respiratory function. BDNF ALS Study Group (Phase III). J Neurol Sci. 1999 Oct 31;169(1-2):13-21. doi: 10.1016/s0022-510x(99)00210-5. PMID 10540002
- [Result] Beghi E, Pupillo E, Bonito V, Buzzi P, Caponnetto C, Chio A, Corbo M, Giannini F, Inghilleri M, Bella VL, Logroscino G, Lorusso L, Lunetta C, Mazzini L, Messina P, Mora G, Perini M, Quadrelli ML, Silani V, Simone IL, Tremolizzo L; Italian ALS Study Group. Randomized double-blind placebo-controlled trial of acetyl-L-carnitine for ALS. Amyotroph Lateral Scler Frontotemporal Degener. 2013 Sep;14(5-6):397-405. doi: 10.3109/21678421.2013.764568. Epub 2013 Feb 19. PMID 23421600
- [Result] Cudkowicz ME, van den Berg LH, Shefner JM, Mitsumoto H, Mora JS, Ludolph A, Hardiman O, Bozik ME, Ingersoll EW, Archibald D, Meyers AL, Dong Y, Farwell WR, Kerr DA; EMPOWER investigators. Dexpramipexole versus placebo for patients with amyotrophic lateral sclerosis (EMPOWER): a randomised, double-blind, phase 3 trial. Lancet Neurol. 2013 Nov;12(11):1059-67. doi: 10.1016/S1474-4422(13)70221-7. Epub 2013 Sep 23. PMID 24067398
- [Result] Dorst J, Cypionka J, Ludolph AC. High-caloric food supplements in the treatment of amyotrophic lateral sclerosis: a prospective interventional study. Amyotroph Lateral Scler Frontotemporal Degener. 2013 Dec;14(7-8):533-6. doi: 10.3109/21678421.2013.823999. Epub 2013 Aug 14. PMID 23944684
- [Result] Lauria G, Campanella A, Filippini G, Martini A, Penza P, Maggi L, Antozzi C, Ciano C, Beretta P, Caldiroli D, Ghelma F, Ferrara G, Ghezzi P, Mantegazza R. Erythropoietin in amyotrophic lateral sclerosis: a pilot, randomized, double-blind, placebo-controlled study of safety and tolerability. Amyotroph Lateral Scler. 2009 Oct-Dec;10(5-6):410-5. doi: 10.3109/17482960902995246. PMID 19922132
- [Result] Miller R, Bradley W, Cudkowicz M, Hubble J, Meininger V, Mitsumoto H, Moore D, Pohlmann H, Sauer D, Silani V, Strong M, Swash M, Vernotica E; TCH346 Study Group. Phase II/III randomized trial of TCH346 in patients with ALS. Neurology. 2007 Aug 21;69(8):776-84. doi: 10.1212/01.wnl.0000269676.07319.09. PMID 17709710
- [Result] Moviglia GA, Moviglia-Brandolino MT, Varela GS, Albanese G, Piccone S, Echegaray G, Martinez G, Blasseti N, Farias J, Farina P, Perusso A, Gaeta CA. Feasibility, safety, and preliminary proof of principles of autologous neural stem cell treatment combined with T-cell vaccination for ALS patients. Cell Transplant. 2012;21 Suppl 1:S57-63. doi: 10.3727/096368912X633770. PMID 22507681
- [Result] Sacca F, Quarantelli M, Rinaldi C, Tucci T, Piro R, Perrotta G, Carotenuto B, Marsili A, Palma V, De Michele G, Brunetti A, Brescia Morra V, Filla A, Salvatore M. A randomized controlled clinical trial of growth hormone in amyotrophic lateral sclerosis: clinical, neuroimaging, and hormonal results. J Neurol. 2012 Jan;259(1):132-8. doi: 10.1007/s00415-011-6146-2. Epub 2011 Jun 25. PMID 21706151
- [Result] Shefner JM, Watson ML, Meng L, Wolff AA; Neals/Cytokinetics STUDY Team. A study to evaluate safety and tolerability of repeated doses of tirasemtiv in patients with amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2013 Dec;14(7-8):574-81. doi: 10.3109/21678421.2013.822517. Epub 2013 Aug 19. PMID 23952636
- [Result] Kaufmann P, Levy G, Montes J, Buchsbaum R, Barsdorf AI, Battista V, Arbing R, Gordon PH, Mitsumoto H, Levin B, Thompson JL; QALS study group. Excellent inter-rater, intra-rater, and telephone-administered reliability of the ALSFRS-R in a multicenter clinical trial. Amyotroph Lateral Scler. 2007 Feb;8(1):42-6. doi: 10.1080/17482960600888156. PMID 17364435
- [Result] Montes J, Levy G, Albert S, Kaufmann P, Buchsbaum R, Gordon PH, Mitsumoto H. Development and evaluation of a self-administered version of the ALSFRS-R. Neurology. 2006 Oct 10;67(7):1294-6. doi: 10.1212/01.wnl.0000238505.22066.fc. PMID 17030772
- [Result] Waitman LR, Aaronson LS, Nadkarni PM, Connolly DW, Campbell JR. The Greater Plains Collaborative: a PCORnet Clinical Research Data Network. J Am Med Inform Assoc. 2014 Jul-Aug;21(4):637-41. doi: 10.1136/amiajnl-2014-002756. Epub 2014 Apr 28. PMID 24778202
- [Result] Mandrioli J, Biguzzi S, Guidi C, Sette E, Terlizzi E, Ravasio A, Casmiro M, Salvi F, Liguori R, Rizzi R, Pietrini V, Borghi A, Rinaldi R, Fini N, Chierici E, Santangelo M, Granieri E, Mussuto V, De Pasqua S, Georgoulopoulou E, Fasano A; ERRALS Group; Ferro S, D'Alessandro R. Heterogeneity in ALSFRS-R decline and survival: a population-based study in Italy. Neurol Sci. 2015 Dec;36(12):2243-52. doi: 10.1007/s10072-015-2343-6. Epub 2015 Jul 24. PMID 26205535
- [Result] Mehta P, Antao V, Kaye W, Sanchez M, Williamson D, Bryan L, Muravov O, Horton K; Division of Toxicology and Human Health Sciences, Agency for Toxic Substances and Disease Registry, Atlanta, Georgia; Centers for Disease Control and Prevention (CDC). Prevalence of amyotrophic lateral sclerosis - United States, 2010-2011. MMWR Suppl. 2014 Jul 25;63(7):1-14. PMID 25054277
- [Result] Gomeni R, Fava M; Pooled Resource Open-Access ALS Clinical Trials Consortium. Amyotrophic lateral sclerosis disease progression model. Amyotroph Lateral Scler Frontotemporal Degener. 2014 Mar;15(1-2):119-29. doi: 10.3109/21678421.2013.838970. Epub 2013 Sep 26. PMID 24070404
- [Result] Gordon PH, Moore DH, Miller RG, Florence JM, Verheijde JL, Doorish C, Hilton JF, Spitalny GM, MacArthur RB, Mitsumoto H, Neville HE, Boylan K, Mozaffar T, Belsh JM, Ravits J, Bedlack RS, Graves MC, McCluskey LF, Barohn RJ, Tandan R; Western ALS Study Group. Efficacy of minocycline in patients with amyotrophic lateral sclerosis: a phase III randomised trial. Lancet Neurol. 2007 Dec;6(12):1045-53. doi: 10.1016/S1474-4422(07)70270-3. Epub 2007 Nov 5. PMID 17980667